CLINICAL TRIAL: NCT05973565
Title: The Effects of a Single Session of Rhythmic Movement Program on Selected Biopsychological Parameters in PD Patients: A Methodological Approach.
Brief Title: The Effects of a Single Session of Rhythmic Movement Program on Selected Biopsychological Parameters in PD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Wolverhampton (Other)
Collaborators: University of Thessaly (Other); National and Kapodistrian University of Athens (Other); Federal University of Rio Grande do Sul (Other); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Matthew Wyon, Prof, University of Wolverhampton
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: YKCK2019
Record Dates: First submitted 2023-05-28; First posted 2023-08-03 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Parkinson Disease; Rhythm
Keywords: musicokinetic education; rhythm; dance; anxiety; gait; walking kinematics; walking kinetics; DLPFC hemodynamics
MeSH Terms: conditions — Parkinson Disease; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Volunteers will be asked to attend three conditions in a randomized order, separated by at least a week of washing out period. Levels of anxiety, kinematic, and DLPFC hemodynamic activity data will be collected before and after the two different interventions, while, on a third occasion, control data will be collected at the same time-points but without any intervention
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Participants will be randomly (randomizer.org) assigned by a researcher blinded to the study either to start with the synchronous intervention or with the asynchronous remote video-based intervention. Two evaluators also blinded to the scope of the study will take all measurements before and after interventions. It will be not possible to blind participants as the delivery of the class will reveal their allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- synchronous learning format (Experimental): Volunteers will be asked to attend synchronous learning format MSK Training. The exercise protocol has a duration of 45 minutes of rhythmic training and includes sections of warming-up, stretching, breathing, movement combinations, a dance sequence and recovery. Each exercise is accompanied with music that provides a clear and predictable rhythm. More specifically, the beat or rhythm of the music is used as a guide for the timing and duration of specific movements, allowing people with PD to coordinate their movements with the music. Simple values are going to be introduced such as whole notes, half notes and quarter notes; clapping and tapping, breathing and sounds. Class will be accompanied by recorded classical piano music, to meet the needs of synchronous learning format and asynchronous remote video-based format. The intensity of the class is moderate approximately 3 MET. The instructor is an experienced dance teacher in musicokinetic education.
  Interventions: Other: Musicokinetic Training
- Asynchronous remote video-based format (Experimental): Volunteers will be asked to attend asynchronous remote video-based format MSK Training.
  The exercise protocol is the same as the synchronous format but delivered via a video-based format
  Interventions: Other: Musicokinetic Training
- Control (No Intervention): Volunteers will not be asked to sit quietly for a 45-minute period

INTERVENTIONS:
Other: Musicokinetic Training — The intervention protocols are either a) synchronous learning format, b) asynchronous remote video- based, and c) control.
  Arms: Asynchronous remote video-based format; synchronous learning format

SUMMARY:
The aim of the present study is to examine the acute effects of a specially designed musicokinetic (MSK) program for patients with Parkinson's disease (PD) on a) anxiety levels b) select kinematic and kinetic parameters, and c) frontal cortex hemodynamic responses, during gait initiation and steady-state walking.

DETAILED DESCRIPTION:
This is a blind cross over randomized control trial (RCT) in which 13 volunteers with PD will attend a 45 min MSK program under the following conditions: a) synchronous learning format, b) asynchronous remote video- based, and c) control conditions. Changes in gait biomechanics and frontal cortex hemodynamic responses will be examined using a 10-camera 3D motion analysis (Vicon T-series, Oxford, UK), and a functional near-infrared spectroscopy (f-NIRS - Portalite, Artinis, NL) system, respectively, while anxiety levels will be evaluated using the Hamilton Anxiety Rating Scale.

ELIGIBILITY:
Inclusion Criteria:

* Hoehn and Yahr (H&Y) Parkinson disease scale I-III
* No restriction on disease duration,
* No restriction on type of drug therapy
* Stable antiparkinsonian medication of at least 6 months
* Data collections will be "on" medication
* No participation to any other exercise program for at least 2 months
* 100% attendance of the session.

Exclusion Criteria:

* Dementia
* Deep brain stimulation,
* Cancer,
* Cardiovascular diseases
* Poor visual capability
* Poor or auditory capability
* Musculoskeletal problems
* No stable antiparkinsonian therapy

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Anxiety | 1-2 hours before the intervention arms and within 2 hours after the completion of the intervention arms
  Hamilton Anxiety rating scale. Scores of 17 or less indicates mild anxiety severity, 18 to 24 indicates mild to moderate anxiety severity, and 25 to 30 indicates a moderate to severe anxiety severity.
Dorsolateral pre-frontal cortex (DLPFC) blood markers during gait | 2 hours before the intervention arms and within 2 hours after the completion of the intervention arms
  A portable fNIRS system (Portalite, Artinis Medical Solutions, Netherlands) will be applied to monitor concentration changes (mM), of O2Hb, HHb and total hemoglobin (tHb) and the difference between O2Hb and HHb [Hbdiff = O2Hb -HHb] of the dorsal lateral prefrontal cortex (DLPFC). To correct for scattering of photons in the tissue, a differential path-length factor (DPF) of 4.0 will be used, for the calculation of absolute concentration changes at a sample frequency of 10Hz. The NIRS probe will be placed in the Brodmann 46 region on the right DLPFC, which has been proposed to be more involved in regulating muscle fatigue and activation. Subsequently, the NIRS probe will be fixed with adhesive tape and a dark elastic bandage around the head to avoid external light and artifacts.
  The O2Hb, HHb and tHb will be used as an indicator of DLPFC total activity, while the Hbdiff (i.e., oxygen supply vs demand) will be used as a marker of oxygenation in the DLPFC.
Gait initiation - balance | 2 hours before the intervention arms and within 2 hours after the completion of the intervention arms
  Using two force plates in line the participant stands on the first, adapting a quite bipedal stance and after a verbal command, starts ambulating forwarding one leg and stepping on the second plate.
  GRFs are calculated from both force plates, to evaluate the balance ability single leg stance (Fy+Fx)
Gait initiation - acceleration | 2 hours before the intervention arms and within 2 hours after the completion of the intervention arms
  Using two force plates in line the participant stands on the first, adapting a quite bipedal stance and after a verbal command, starts ambulating forwarding one leg and stepping on the second plate.
  GRFs are calculated from both force plates, to evaluate foot clear force (FZ) respectively (leg .1)
Walking kinematic parameters - stride length | 2 hours before the intervention arms and within 2 hours after the completion of the intervention arms
  Ground reaction force (GRF) data captured at 1000 Hz for the right and left leg by the force platforms will be synchronized with the kinematic data obtained by the Vicon motion analysis system at 1000 Hz. Kinematic data will focus on stride length and time and shoulder-pelvis association.
Walking kinematic parameters - shoulder-pelvis association | 2 hours before the intervention arms and within 2 hours after the completion of the intervention arms
  Kinematic data obtained by the Vicon motion analysis system at 1000 Hz will focus on shoulder-pelvis association.
Walking kinematic parameters - gait velocity | 2 hours before the intervention arms and within 2 hours after the completion of the intervention arms
  Kinematic data obtained by the Vicon motion analysis system at 1000 Hz and will focus on gait velocity.
Walking kinetic parameters - medio-lateral ground reaction forces | 2 hours before the intervention arms and within 2 hours after the completion of the intervention arms
  GRFs are calculated from both force plates, to evaluate the medio-lateral movement during the stance phase of walking (Fy+Fx)
Walking kinetic parameters- foot strike | 2 hours before the intervention arms and within 2 hours after the completion of the intervention arms
  GRFs are calculated from both force plates, to evaluate the strike forces during landing (Fz)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wolverhampton, Walsall, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No